CLINICAL TRIAL: NCT03347955
Title: Transplantation of Embryonic Dopamine Neurons for Treatment of Parkinson's Disease: Double-blind Placebo Surgery Trial
Brief Title: Double-blind Placebo Surgery Trial for Treatment of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Denver (Other)
Responsible Party: Principal Investigator, Cynthia McRae, PhD, Research Professor, University of Denver
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R29NS032009-05 (NIH)
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Parkinson Disease; Surgery
Keywords: placebo effect
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: In this double-blind study, 20 participants were randomly assigned to the treatment group and 20 to the sham surgery group with the blind being maintained for 12 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All of the above were "masked." Only the neurosurgeon (Dr. Breeze) who did the implant and the person in charge of random assignment were aware of which participant received which treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural implantation group (Experimental): Human embryonic dopamine neurons were implanted into brains of half the randomized participants (n = 20). Participants were evaluated at baseline, 4, 8, and 12 months after surgery.
  Interventions: Procedure: Neural implantation group
- Sham Surgery group (Sham Comparator): This group (n = 20) received sham surgery with a steel frame affixed to their heads and four burr holes drilled into their foreheads without crossing the blood/brain barrier. Participants were assessed at baseline, 4, 8, and 12 months after surgery.
  Interventions: Procedure: Sham surgery

INTERVENTIONS:
Procedure: Neural implantation group — Cultured mesencephalic tissue from four embryos was implanted into the putamen bilaterally for those receiving the implant
  Arms: Neural implantation group
Procedure: Sham surgery — Steel frame affixed to head and four burr holes drilled into forehead of sham surgery patients
  Arms: Sham Surgery group

SUMMARY:
A double-blind sham surgery-controlled trial was developed to determine the effectiveness of implantation of human embryonic dopamine neurons into the putamen of patients with advanced Parkinson's disease (PD), with half the patients receiving the implant (n = 20) and half receiving sham surgery (n = 20). The blind was maintained for 12 months before participants were told which surgery they received, at which time those receiving sham surgery could request the implant surgery.

DETAILED DESCRIPTION:
A double-blind sham surgery-controlled trial was conducted to determine the effectiveness of implantation of human embryonic dopamine neurons into the putamen of patients with advanced Parkinson's disease (PD), with half the patients receiving the implant (n = 20) and half receiving sham surgery (n = 20). The goals were to determine whether the cells survived and led to improvement of symptoms, and to examine the effect of age on results of the implantation. Quality of life of participants and care partners was also examined at each of the assessment periods (baseline, 4, 8 and 12 months). The blind was maintained for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease (PD) for more than 7 years, improvement in response to levodopa, Positive Emission Tomography scan compatible with presence of PD, improvement of at least 33% on UPDRS after first morning dose of levodopa

Exclusion Criteria:

* Mini-mental status exam score of less than 24, hallucinations during levodopa therapy, epilepsy, previous brain surgery, severe depression, another neurologic disorder, cardiovascular disease, and medical contraindication of surgery

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1994-11 (Actual); Primary Completion 1999-02 (Actual); Study Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Global Rating Scale | Same scale was administered 7 days after surgery and prior to follow-up visits at Columbia at 4, 8, and 12 months after surgery and before the blind was lifted.
  one item scale where participants marked their answer on a scale ranging from -3 (much worse since surgery) to 0 (no change) to +3 (much improved since surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia McRae, PhD, Principal Investigator — University of Denver; Stanley Fahn, MD, Study Chair — Neurological Institute, Columbia University; Curt Freed, MD, Study Director — University of Colorado Health Sciences
Locations (1):
- Morgridge College of Education, University of Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McRae C, Cherin E, Yamazaki TG, Diem G, Vo AH, Russell D, Ellgring JH, Fahn S, Greene P, Dillon S, Winfield H, Bjugstad KB, Freed CR. Effects of perceived treatment on quality of life and medical outcomes in a double-blind placebo surgery trial. Arch Gen Psychiatry. 2004 Apr;61(4):412-20. doi: 10.1001/archpsyc.61.4.412. PMID 15066900
- [Result] Freed CR, Greene PE, Breeze RE, Tsai WY, DuMouchel W, Kao R, Dillon S, Winfield H, Culver S, Trojanowski JQ, Eidelberg D, Fahn S. Transplantation of embryonic dopamine neurons for severe Parkinson's disease. N Engl J Med. 2001 Mar 8;344(10):710-9. doi: 10.1056/NEJM200103083441002. PMID 11236774
- See also: Quality of life report on double-blind fetal transplant surgery for treatment of Parkinsons disease — https://www.ncbi.nlm.nih.gov/pubmed?term=%22Archives+of+general+psychiatry%22%5BJour%5D+AND+2004%5Bpdat%5D+AND+McRae+C%5Bauthor%5D&cmd=detailssearch
- See also: Neurological and medical results of double-blind fetal transplant surgery as treatment for Parkinson's disease — https://www.ncbi.nlm.nih.gov/pubmed?term=%22The+New+England+journal+of+medicine%22%5BJour%5D+AND+344%5Bvolume%5D+AND+2001%5Bpdat%5D+AND+Freed%5Bfirst+author%5D+AND+Transplantation&TransSchema=title&cmd=detailssearch